CLINICAL TRIAL: NCT02806817
Title: ME-344 in Early HER2-negative Breast Cancer With Antiangiogenic-induced Mitochondrial Metabolism: a Phase 0 Trial
Brief Title: ME-344 in Early HER2-negative Breast Cancer With Antiangiogenic-induced Mitochondrial Metabolism
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centro Nacional de Investigaciones Oncologicas CARLOS III (Other)
Collaborators: Fundacion CRIS de Investigación para Vencer el Cáncer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CNIO-BR-009; 2015-005457-12 (EudraCT Number)
Record Dates: First submitted 2016-05-20; First posted 2016-06-21 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast; Early-Stage Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — ME-344; Bevacizumab; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bevacizumab + ME-344 (Experimental): Bevacizumab single dose (15 mg/kg infused IV) on day 1. ME-344 will be administered at 10 mg/kg infused IV over 30 minutes on days 8, 15 and 22 (arm 1).
  ME-344 will be suspended in 250 mL sterile saline.
  Interventions: Drug: ME-344; Drug: Bevacizumab
- Bevacizumab + normal saline (Placebo Comparator): Bevacizumab single dose (15 mg/kg infused IV) on day 1. Placebo: will be administered normal saline 250 mL infused IV over 30 minutes on days 8, 15 and 22 (arm 2).
  Interventions: Drug: Bevacizumab; Other: Normal saline

INTERVENTIONS:
Drug: ME-344 — ME-344 is a synthetic small molecule mitochondrial inhibitor based on the isoflavan ring structure. ME-344 is a chiral compound, and is manufactured predominantly as a single stereoisomer that is dextrorotatory. As a stereoisomeric drug with two chiral centers, ME-344 is one of four potential stereoisomers. The current manufacturing process produces a racemic mixture of two of those stereoisomers, which are enantiomers, and ME-344 is separated from the levorotatory enantiomer by chromatography in the final step.
  Other Names: small molecule mitochondrial inhibitor
  Arms: Bevacizumab + ME-344
Drug: Bevacizumab — Bevacizumab is a recombinant humanized monoclonal antibody that blocks angiogenesis by inhibiting vascular endothelial growth factor A (VEGF-A)
  Other Names: Avastin
Other: Normal saline — Use saline as placebo
  Arms: Bevacizumab + normal saline

SUMMARY:
Prospective, randomized, open label, two arms,, phase 0 clinical trial. HER2-negative breast cancer patients recently diagnosed will be screened for trial participation.

A biopsy will be scheduled the week prior to or the same day as the FDG PET. Paraffin-embedded tumor samples will be used to evaluate the stainings of Ki67, cleaved caspase-3 and microvessels, and frozen tumor samples will be used to evaluate SDH staining.

The FDG-PET will be followed by the bevacizumab dose (15 mg/kg IV, single dose). After one week, the PET will be repeated in order to detect the patients that have experienced FDG uptake decay.

Right after, treatment with ME-344 (arm 1) or no treatment (arm 2) will start. ME-344 will be administered at 10 mg/kg on day 8, 15 and 22. Surgery will be performed on day 28 (thus, 4 weeks after the bevacizumab dose, which is considered a safe window for antiangiogenics).

Fragments of the surgical specimen will be collected. Paraffin-embedded tumor sample will be used to repeat (and compare) the stainings of Ki67, cleaved caspase-3 and microvessels, and frozen tumor sample will be used to repeat (and compare) SDH staining.

Patients will come off trial in case of consent withdrawal, unequivocal disease progression is observed, unacceptable toxicity occurs, or in case of intercurrent disease or any other condition deemed incompatible with continuation in the clinical trial by the investigator.

DETAILED DESCRIPTION:
Antiangiogenic agents are the most widely used biologic agents in oncology and are approved by the Food and Drug Administration (FDA) for use against many different malignancies based on the results of several randomized phase III trials. However, acquired resistance to antiangiogenics is a major problem in cancer therapeutics.

Some signaling nodes have been implicated in therapeutic resistance in preclinical studies. However, a global tumor-reprogramming interrogation based on changes in the delivery of oxygen and nutrients has not been undertaken. The findings link acquired resistance to a powerful anticancer drug class with aberrant cancer metabolism. Under selective pressure, tumor plasticity allows sustained tumor growth in the long term despite exposure to antiangiogenic TKIs, and it renders mitochondrial metabolism essential for survival When one energy source (glycolysis) is pharmacologically limited, the tumors become vulnerable to the inhibition of the other (mitochondrial metabolism). Pharmacological blockers of the nutritional stress regulators can abrogate mitochondrial respiration and tumor growth in this situation, which the investigators have termed "metabolic synthetic lethality".

The investigators hypothesized that in cases in which antiangiogenics lead to hypoxia normalization, chronic high-rate glycolysis is offset and tumors might switch to an alternative metabolic source. If this source is essential for tumor survival, it would open a therapeutic opportunity.

The administration of ME-344 in animals where antiangiogenics have induced a mitochondrial phenotype seems promising. The investigators aim to extend these observations in humans. However, several questions remain, prior to launch a large trial:

* Which percentage of patients experience a mitochondrial shift when exposed to a given antiangiogenic.
* In case this happens, whether it is possible to trace this response accurately.
* What is the benefit of adding ME-344 in those cases showing the mitochondrial shift, and what is the benefit, if any, of adding it in the remainder cases.

For that purpose, investigators will conduct a pilot randomized phase 0 trial, where a cohort of patients will be treated with a single bevacizumab dose prior to surgery and a second cohort with bevacizumab plus ME-344.

The purpose of this clinical trial is to evaluate if the addition of ME-344 to antiangiogenic agents in the cases where the mitochondrial phenotype has been induced will enhance antitumor activity.

ELIGIBILITY:
Inclusion Criteria:

1. Women older than 18 year-old.
2. Treatment-naïve diagnosed early (stage I-III) HER2-negative (histologically confirmed) breast cancer not candidates for neoadjuvant therapy.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Signed informed consent obtained from the subject prior to performing any protocol-related procedures.
5. Negative pregnancy test, or confirmed menopause.
6. Adequate organ function, according to the following parameters:

   * Haemoglobin ≥ 9.0 g/dL.
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 / mm3).
   * Platelet count ≥ 100 x 109/L (>100000 / mm3).
   * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal.
   * Serum creatinine < 1.5 x institutional upper limit of normal (ULN).
7. Cardiac ejection fraction above 45%.
8. Life expectancy superior to 6 months.
9. Willingness to undergo trial procedures.

Exclusion Criteria:

1. Neuropathy of any kind.
2. Diabetes mellitus.
3. Presence of intercurrent uncontrolled diseases, including untreated hypertension.
4. Participation in another clinical study with an investigational product during the last 4 weeks.
5. Patients with presence of concurrent or active malignant disease (other than disease under study) within the last 12 months with the exception of adequately treated in situ carcinomas, basal or squamous cell carcinoma, or nonmelanomatous skin cancer.
6. Female subjects who are pregnant, breast-feeding or of reproductive potential who are not employing an effective method of birth control.
7. Uncontrolled infection or systemic disease.
8. Clinically significant cardiac disease not well controlled with medication (e.g., congestive heart failure, symptomatic coronary artery disease e.g. angina, and cardiac arrhythmias) or myocardial infarction within the last 12 months.
9. No concurrent systemic chemotherapy or biologic therapy is allowed.
10. Known hypersensitivity to any components of ME-344 or bevacizumab.
11. Known human immunodeficiency virus (HIV) or Hepatitis B or C (active, previously treated or both).
12. History of solid organ transplantation.
13. Psychiatric disorder or social or geographic situation that would preclude study participation.
14. Inability to comply with the study and follow-up procedures (e.g. tumor biopsies).
15. Any other condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Reduction of FDG uptake | 1 month
  Mitochondrial switch changes from baseline
SDH (succinate dehydrogenase) levels staining | 1 month
  Mitochondrial switch changes from baseline: glucolisis and studies microvasculature

SECONDARY OUTCOMES:
Toxicity profile: Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | 8 weeks
  All toxicities will be graded according to NCI CTCAE v4.03
Ki67 changes | From day 1 to day 8
  Antitumor activity: Ki67 changes
Cleaved caspase-3 changes | From day 1 to day 8
  Antitumor activity: Cleaved caspase-3 changes

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - H. Arnau de Vilanova Lleida, Lleida
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Clínica Quirón, Madrid

IPD SHARING:
Plan to Share IPD: Undecided